CLINICAL TRIAL: NCT06680635
Title: Role of Microbiota, Inflammation and Oxidative Stress in the Pathophysiology of Obesity: Therapeutic Potential of Citrus Flavonoids
Brief Title: Effect of Citrus Flavonoids on Obesity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celia Bañuls (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Celia Bañuls, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI21/01160
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Obesity Adult Onset; Diabetes Mellitus Type 2
Keywords: Polyphenols; Microbiota; Inflammation; Oxidative stress; Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flavonoid-enriched juice and low-calorie diet for obese patients (Active Comparator): Subjects will receive nutritional intervention by a registered dietician and a flavonoid-enriched juice supplement for 8 weeks. The dietary intervention consists of healthy dietary recommendations and hypocaloric diet if necessary (overweight, obesity).
  Interventions: Dietary Supplement: Flavonoid-enriched juice and a low-calorie diet
- Pacebo juice and low-calorie diet for obese patients (Placebo Comparator): Subjects will receive nutritional intervention by a registered dietitian and a placebo in the form of juice for 8 weeks. The dietary intervention consists of healthy dietary recommendations and hypocaloric diet if necessary (overweight, obesity).
  Interventions: Dietary Supplement: Food supplement: placebo juice and a low calorie diet

INTERVENTIONS:
Dietary Supplement: Flavonoid-enriched juice and a low-calorie diet — Orange juice enriched in flavonoids (14%: nobiletin, sinensetin, tangeretin) (200 ml/day) and low calorie diet
  Arms: Flavonoid-enriched juice and low-calorie diet for obese patients
Dietary Supplement: Food supplement: placebo juice and a low calorie diet — Placebo juice (200 ml/day) and a low calorie diet
  Arms: Pacebo juice and low-calorie diet for obese patients

SUMMARY:
The aim of this study is to evaluate whether the intake of a functional juice enriched in citrus polymethoxylated flavonoids is able to improve the glycaemic profile and insulin resistance of obese patients by reversing the associated oxidative and inflammatory stress, as well as the differential alteration of the intestinal microbiota. To achieve this, a prospective, randomised, double-blind, placebo- controlled, clinical-baseline intervention study will be conducted in obese patients (BMI=30-40 kg/m2) with type 2 diabetes (DM2) (n=40) and obese patients without alterations in carbohydrate metabolism (n=40). Each of these groups will be randomly divided into 2 subgroups (n=20), one of which will receive polymethoxyflavonoid-enriched orange juice (14%: nobiletin, sinensetin, tangeretin) (200 ml/ day) and the other group will receive the corresponding placebo juice for 8 weeks. In addition, all of them will receive a hypocaloric diet. Anthropometric parameters, body composition and nutritional status will be assessed, cardiovascular risk factors and comorbidities will be studied (HT, SAHS, dyslipidaemia, insulin resistance), oxidative stress parameters will be compared (total and mitochondrial ROS production, mitochondrial membrane potential, glutathione levels by static cytometry and mitochondrial respiration rate by Seahorse flow analyser), antioxidant enzymes (SOD, GPx) and molecular oxidation products (Carbonyl proteins and 8-oxo-dG, LDLox) and LPS by ELISA techniques, inflammatory parameters (IL6, TNFa, IL1b, adiponectin, PAI-1, IL10) by Luminex XMAP technology in serum. Metabolomic analysis will also be performed in plasma (NMR spectroscopy and PLS-DA), and the content and diversity of the gut microbiota (16S rRNA amplicons, and direct metagenomic sequencing, with Illumina MiSeq technology) will be assessed in faeces, before and after the dietary intervention. Individualised dietary follow-up and assessment of subjects' quality of life will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* patients with a BMI of 30 -40 kg/m2, between 18 and 65 years of age.
* Obesity of more than five years' duration
* Patients will maintain a stable weight (±2 kg) during the 3 months prior to the study.

Exclusion Criteria:

* Patients with acute or chronic inflammatory diseases and established liver and kidney failure (based on transaminase levels ±2 SD of the mean and estimated glomerular filtration rate using the CKD-EPI formula >60), neoplastic diseases and secondary causes of obesity (hypothyroidism, Cushing's syndrome), use of drugs that may influence inflammatory status or insulin sensitivity (NSAIDs, corticosteroids, anti-TNFα), treatment with insulin or GLP1 inhibitors, type 1 diabetes, morbid obesity (BMI>40 kg/m2), hypertriglyceridaemia (> 400 mg/dl), fructose intolerance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
To evaluate insulin resistance index | 5 years
  Evaluate if there is an improvement in insulin resistance levels after the intervention depending on the intake of a flavonoid-enriched juice or its corresponding placebo for 6 weeks, in obese patients without alterations in carbohydrate metabolism and obese patients with type 2 diabetes (DM2).
  HOMA-IR will be used. Participants will be considered to have achieved an improvement in insulin resistance levels if they normalize its value (normality values defined between 0 and 3.8 units).
Analyze the significant differences between metabolomic profile before and after the dietetic intervention, and between both groups (flavonoid-enriched juice vs placebo).. | 5 years
  NMR spectra will be used to obtain spectra from serum samples from the cohort. In order to evaluate if there will be significant differences after the dietetic intervention, a PLS-DA model for discrimination between basal and post intervention levels will be performed. Scores plots will be calculated with a 95% confidence interval.

SECONDARY OUTCOMES:
Assess significant changes in body fat mass percentage after the dietetic intervention. | 5 years
  Percentage of body fat mass will be measured by bioelectrical impedance. It is considered to be high when ≥25% in men and ≥30% in women. A significant improvement will be considered when notable differences are observed in the mean values between groups (flavonoid-enriched juice vs. placebo) measured through p-value (<0.05) with a 95% confidence interval.
To assess significant changes in triglycerides before and after the use of flavonoid-enriched juice and its placebo in the same groups of patients. | 5 years
  Participants will be considered to have achieved an improvement in plasmatic triglycerides level if they normalize its value (normality values defined between 0 and 150mg/dL).
To evaluate the composition and diversity of gut microbiota | 5 years
  To evaluate the diversity of gut microbiota in faeces (measured by alpha-diversity) before and after the use of a flavonoid-enriched juice and its placebo in the same groups of patients.
  To asses the differences in alpha-diversity of the intestinal microbiota in both groups, it will be evaluated whether there are significant differences between the Shannon indices of the two groups. The results are interpreted as follows: values less than 2 are considered low in diversity and values greater than 3 are high in species diversity.
To identify serum biomarkers using a metabolomic approach | 5 years
  To identify serum biomarkers using a metabolomic approach before and after intervention with flavonoid-enriched juice or placebo in the same groups of patients. NMR spectra will be used to obtain spectra from serum samples from the cohort. In order to evaluate if there will be significant differences after the dietetic intervention (according to the flavonoid-enriched juice or placebo intake), a PLS-DA model for discrimination between basal and post intervention levels will be performed. Scores plots will be calculated with a 95% confidence interval.
Evaluate significant changes in % of weight loss after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
To assess significant changes in LDLc before and after the use of flavonoid-enriched juice and its placebo in the same groups of patients. | 5 years
  Participants will be considered to have achieved an improvement in serum cLDL levels if they normalize its value (normality values defined between 0 and 130mg/dL).
To assess significant changes in HDLc before and after the use of flavonoid-enriched juice and its placebo in the same groups of patients. | 5 years
  Participants will be considered to have achieved an improvement in serum cHDL levels if they normalize its value (normality values defined between 45 and 70mg/dL in women, and 40 to 70mg/dL in men).
Evaluate significant changes in high-sensitivity C-reactive protein (hs-CRP) after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  Participants will be considered to have achieved an improvement in high-sensitivity C-reactive protein levels if they normalize its value (normality values defined between 0 and 1.69mg/dl).
Assess significant changes in C3 protein after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  Participants will be considered to have achieved an improvement in C3 protein if they normalize its value (normality values defined between 81 and 157mg/dl).
Evaluate significant changes in plasmatic homocysteine as a inflammatory parameter after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  Participants will be considered to have achieved an improvement in plasmatic homocysteine if they normalize its value (normality values defined between 5 and 15µmol/L).
Assess significant changes in interleukin 1-beta (IL-1B) levels as a pro-inflammatory molecule after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  IL-1B levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate significant changes in interleukin 6 (IL-6) levels as a pro-inflammatory molecule after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  IL-6 levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess significant changes in tumor necrosis factor alpha (TNF-alpha) levels as a pro-inflammatory molecule after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  TNF-alpha levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate significant changes in superoxide dismutase (SOD) levels as a pro-inflammatory molecule after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  Superoxide dismutase levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate significant changes in ROS levels after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  Total ROS levels will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess significant improvements in glutathione levels after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  Total glutathione levels will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess significant improvements in total free radicals and superoxide levels after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  Total free radicals and superoxide content will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Evaluate significant improvements in mitochondrial ROS production after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  Mitochondrial ROS production will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Analyze significant improvements in mitochondrial membrane potential after the dietetic intervention in both groups (flavonoid-enriched juice vs placebo) after the dietary intervention. | 5 years
  Mitochondrial membrane potential will be assessed by a flow cytometry assay in PBMCs. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Locations (1):
- FISABIO, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No